CLINICAL TRIAL: NCT02423551
Title: Effects of Meal, Ready-to-Eat (MRE) Consumption on Gut Health
Brief Title: MRE Consumption and Gut Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Philip Karl, Research Dietitian, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-12HC
Record Dates: First submitted 2015-04-14; First posted 2015-04-22 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Gastrointestinal Tract
Keywords: Gut microbiota; Intestinal permeability; Gut barrier integrity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual diet
- MRE (Experimental): MRE consumption
  Interventions: Other: MRE

INTERVENTIONS:
Other: MRE — MRE consumption
  Arms: MRE

SUMMARY:
The objective of this study is to determine the impact of consuming MREs as the sole source of subsistence for 21 days on gut bacteria community composition and gut health. Up to 80 free-living adults will be randomized to consume their usual diet or only MREs for 21 consecutive days. MREs will be provided by the Military Nutrition Division, US Army Research Institute of Environmental Medicine (USARIEM). Fecal, urine and blood samples will be collected periodically before, during and after the intervention to measure gut barrier integrity, gut bacteria community composition, and markers of gut health, inflammation, and nutritional status.

ELIGIBILITY:
Inclusion Criteria:

* BMI </= 30

Exclusion Criteria:

* Use of antiobiotcs within 3 months of study participation
* Use of pro- or prebiotic supplements within 2 weeks of study participation
* Vegetarian diets
* Use of laxatives, stool softeners, or anti-diarrheal medications at least once a week.
* Fewer than 4 bowel movements, on average, per week
* History of gastrointestinal disease
* Colonoscopy within 3 months of study participation
* Food allergies or aversions or other issues with foods that would preclude MRE consumption, including gluten, milk, nuts, or eggs.
* Use non-steroidal anti-inflammatory medications (NSAIDs) or antihistamine prescribed by a physician or clinician, or unwillingness to discontinue the use of these substances during the study.
* Actively trying to lose weight
* Pregnant or lactating
* Recent blood donation

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in gut barrier integrity | Baseline to 10 days, 21 days and 31 days
  Urine excretion of saccharide probes; circulating zonulin, intestinal fatty acid binding protein, claudin-3, lipopolysaccharide and GLP2 concentrations

SECONDARY OUTCOMES:
Change in gut microbiota composition | Baseline to 10 days, 21 days and 31 days
  16S rRNA gene sequencing
Change in C-reactive protein concentrations | Baseline to 10 days, 21 days and 31 days
  Serum C-reactive protein
Change in TNF-alpha concentrations | Baseline to 10 days, 21 days and 31 days
  Serum TNF-alpha
Change in interleukin-6 concentrations | Baseline to 10 days, 21 days and 31 days
  Serum IL-6
Change in lipopolysaccharide concentrations | Baseline to 10 days, 21 days and 31 days
  Plasma LPS
Change in iron status | Baseline to 10 days, 21 days and 31 days
  Blood ferritin, soluble transferrin receptor, hemoglobin, hematocrit
Change in vitamin D status | Baseline to 10 days, 21 days and 31 days
  Blood 25-hydroxyvitamin D, 1,25-dihydroxyvitamin D, parathyroid hormone
Change in B-vitamin status | Baseline to 10 days, 21 days and 31 days
  Blood folate, vitamin B12, homocysteine
Change in nutritional status | Baseline to 10 days, 21 days and 31 days
  Blood prealbumin
Change in calcium absorption | Baseline to 10 days, 21 days and 31 days
  Urine calcium
Change in zinc status | Baseline to 10 days, 21 days and 31 days
  Blood zinc, zinc receptor expression

CONTACTS AND LOCATIONS:
Locations (1):
- USARIEM, Natick, Massachusetts, United States

REFERENCES:
- [Derived] Karl JP, Armstrong NJ, Player RA, Rood JC, Soares JW, McClung HL. The Fecal Metabolome Links Diet Composition, Foacidic positive ion conditions, chromatographicallyod Processing, and the Gut Microbiota to Gastrointestinal Health in a Randomized Trial of Adults Consuming a Processed Diet. J Nutr. 2022 Nov;152(11):2343-2357. doi: 10.1093/jn/nxac161. Epub 2022 Jul 26. PMID 36774101
- [Derived] Pantoja-Feliciano IG, Karl JP, Perisin M, Doherty LA, McClung HL, Armstrong NJ, Renberg R, Racicot K, Branck T, Arcidiacono S, Soares JW. In vitro gut microbiome response to carbohydrate supplementation is acutely affected by a sudden change in diet. BMC Microbiol. 2023 Jan 28;23(1):32. doi: 10.1186/s12866-023-02776-2. PMID 36707764
- [Derived] McClung HL, Armstrong NJ, Hennigar SR, Staab JS, Montain SJ, Karl JP. Randomized Trial Comparing Consumption of Military Rations to Usual Intake for 21 Consecutive Days: Nutrient Adequacy and Indicators of Health Status. J Acad Nutr Diet. 2020 Nov;120(11):1791-1804. doi: 10.1016/j.jand.2020.06.018. Epub 2020 Aug 19. PMID 32828737